CLINICAL TRIAL: NCT06755242
Title: An Open-label, Multicenter, Phase I Clinical Study to Evaluate the Safety, Tolerability, Pharmacokinetics Characteristics or Preliminary Efficacy and Antitumor Activity of GNC-077 Multi-specific Antibody Injection in Patients With Locally Advanced or Metastatic Gastrointestinal Tumors and Other Solid Tumors
Brief Title: A Study of GNC-077 in Patients With Locally Advanced or Metastatic Gastrointestinal Tumors and Other Solid Tumors
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Sichuan Baili Pharmaceutical Co., Ltd. (Industry)
Collaborators: Baili-Bio (Chengdu) Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GNC-077-103
Record Dates: First submitted 2024-12-25; First posted 2025-01-01 (Actual); Last update posted 2025-01-01 (Actual); Status verified 2024-12

CONDITIONS: Gastrointestinal Tumors; Solid Tumor
MeSH Terms: conditions — Digestive System Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- GNC-077 (Experimental): Participants receive GNC-077 as intravenous infusion for the first cycle (3 weeks). Participants with clinical benefit could receive additional treatment for more cycles. The administration will be terminated because of disease progression or intolerable toxicity occurring or other reasons.
  Interventions: Drug: GNC-077

INTERVENTIONS:
Drug: GNC-077 — Administration by intravenous infusion for a cycle of 3 weeks.

SUMMARY:
This study is an open-label, multicenter, dose-escalation and cohort expansion phase I clinical study to evaluate the safety, tolerability, pharmacokinetics characteristics or preliminary efficacy and antitumor activity in patients with locally advanced or metastatic gastrointestinal tumors and other solid tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Able to understand the informed consent form, voluntarily participate in and sign the informed consent form;
2. Gender is not limited;
3. Age: ≥18 years old and ≤75 years old (phase Ia); ≥18 years old (phase Ib);
4. Patients with locally advanced or metastatic gastrointestinal tumors and other solid tumors confirmed by histopathology and/or cytology who failed standard treatment;
5. Must have at least one measurable lesion that meets the RECIST v1.1 definition;
6. Have archived primary or recurrent tumor tissue specimens that can be submitted for central review;
7. ECOG ≤1;
8. The expected survival time as judged by the investigators was ≥3 months;
9. Bone marrow function, renal function and liver function need to meet the requirements;
10. Coagulation function: fibrinogen ≥1.5 g/L; Activated partial thromboplastin time (APTT) ≤1.5×ULN; Prothrombin time (PT) ≤1.5×ULN;
11. Fertile female subjects or male subjects with fertile partners must use highly effective contraception from 7 days before the first dose until 12 weeks after the last dose. Female subjects of childbearing potential must have a negative serum pregnancy test within 7 days before the first dose;
12. Subjects were able and willing to comply with protocol-specified visits, treatment plans, laboratory tests, and other study-related procedures.

Exclusion Criteria:

1. Chemotherapy, biological therapy, immunotherapy and other anti-tumor therapies have been used within 4 weeks or 5 half-lives before the first dose; Mitomycin and nitrosoureas were administered within 6 weeks before the first dose; Oral drugs such as fluorouracil;
2. Patients with active infection requiring intravenous antibiotics that had not been completed more than 1 week before enrollment, with the exception of prophylactic antibiotics for puncture or biopsy;
3. Positive human immunodeficiency virus antibody, active tuberculosis, active hepatitis B virus infection or hepatitis C virus infection;
4. Toxicity from prior antineoplastic therapy is not reduced to grade I as defined in CTCAE, version 5.0;
5. Patients at risk for active autoimmune disease or with a history of autoimmune disease may have central nervous system involvement;
6. Pulmonary disease defined as ≥ grade 3 according to NCI-CTCAE v5.0; A history of ILD requiring steroid therapy, or current ILD or grade ≥2 radiation pneumonitis;
7. Patients with previous allogeneic hematopoietic stem cell transplantation or organ transplantation;
8. Had a history of severe cardiovascular and cerebrovascular diseases;
9. Patients with or with unstable thrombotic events such as deep vein thrombosis, arterial thrombosis and pulmonary embolism within 6 months before screening;
10. Brain parenchymal metastases and/or meningeal metastases or spinal cord compression, excluding stable and asymptomatic brain parenchymal metastases;
11. Patients with massive or symptomatic effusions or poorly controlled effusions;
12. Imaging examination showed that the tumor had invaded or wrapped around the chest, neck, pharynx and other large arteries;
13. Subjects with clinically significant bleeding or significant bleeding tendency within the previous 4 weeks were screened;
14. Complicated with other malignant tumors within 3 years before the first administration;
15. Poorly controlled hypertension (systolic blood pressure > 150 mmHg or diastolic blood pressure > 100 mmHg);
16. Diabetic patients with poor glycemic control;
17. Patients with a history of allergy to recombinant humanized antibodies or to any of the excipients of GNC-077;
18. Who had participated in a clinical trial of an unmarketed drug within 4 weeks before the trial dose;
19. Had received a live vaccine within 4 weeks before the trial dose;
20. Other circumstances that the investigator deemed inappropriate for participation in the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-01 (Estimated); Primary Completion 2027-06 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Phase Ia: Dose limiting toxicity (DLT) | Up to 21 days after the first dose
  DLTs are assessed according to NCI-CTCAE v5.0 during the first cycle and defined as occurrence of any of the toxicities in DLT definition if judged by the investigator to be possibly, probably or definitely related to study drug administration.
Phase Ia: Maximum tolerated dose (MTD) | Up to 21 days after the first dose
  MTD is defined as the highest dose level at which no more than 1 in 6 participants experienced a DLT during the first cycle.
Phase Ia: Treatment-Emergent Adverse Event (TEAE) | Up to approximately 24 months
  TEAE is defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally emerging, or any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a pre-existing condition during the treatment of GNC-077 . The type, frequency and severity of TEAE will be evaluated during the treatment of GNC-077.
Phase Ib: Recommended Phase II Dose (RP2D) | Up to approximately 24 months
  The RP2D is defined as the dose level chosen by the sponsor (in consultation with the investigators) for phase II study, based on safety, tolerability, efficacy, PK, and PD data collected during the dose escalation study of GNC-077.

SECONDARY OUTCOMES:
Cmax | Up to approximately 24 months
  Maximum serum concentration (Cmax) of GNC-077 will be investigated.
Tmax | Up to approximately 24 months
  Time to maximum serum concentration (Tmax) of GNC-077 will be investigated.
AUC0-inf | Up to approximately 24 months
  AUC0-inf is defined as area under the concentration-time curve from 0 to inf.
AUC0-t | Up to approximately 24 months
  AUC0-t is defined as area under the serum concentration-time curve from time 0 to the time of the last measurable concentration.
CL (Clearance) | Up to approximately 24 months
  CL in the serum of GNC-077 per unit of time will be investigated.
T1/2 | Up to approximately 24 months
  Half-life (T1/2) of GNC-077 will be investigated.
ADA (anti-drug antibody) | Up to approximately 24 months
  Frequency of anti-GNC-077 antibody (ADA) will be investigated.
Objective Response Rate (ORR) | Up to approximately 24 months
  ORR is defined as the percentage of participants, who has a CR (disappearance of all target lesions) or PR (at least a 30% decrease in the sum of diameters of target lesions). The percentage of participants who experiences a confirmed CR or PR is according to RECIST 1.1.
Progression-free survival (PFS) | Up to approximately 24 months
  The PFS is defined as the time from the participant's first dose of GNC-077 to the first date of either disease progression or death, whichever occurs first.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Cancer Hospital, Beijing, Beijing Municipality, China